CLINICAL TRIAL: NCT06197425
Title: Phase III Multicentric, Open-label, Randomized Study to Investigate the Efficacy of Chemotherapy in Patients With Positive ctDNA After Surgery and Adjuvant Chemotherapy for a Stage III Colorectal Cancer (PRODIGE 88)
Brief Title: Investigate the Efficacy of Chemotherapy in Patients With Positive ctDNA After Surgery and Adjuvant Chemotherapy for a Stage III Colorectal Cancer
Acronym: CIRCULATE PAC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEPAGE PHRCK 2022
Record Dates: First submitted 2023-12-22; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Colon or Upper Rectum Adenocarcinoma
MeSH Terms: interventions — Surveys and Questionnaires; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chemotherapy by FOLFIRI (Experimental)
  Interventions: Drug: "FOLFIRI" cures; Biological: BIOLOGICAL ASSESSMENT; Other: Questionnaires; Other: Thoracic-abdomino-pelvic scan or MRI
- Chemotherapy by Trifluridine tipiracil (Experimental)
  Interventions: Drug: Trifluridine cures; Biological: BIOLOGICAL ASSESSMENT; Other: Questionnaires; Other: Thoracic-abdomino-pelvic scan or MRI
- Surveillance inside the trial/control arm (Active Comparator)
  Interventions: Biological: BIOLOGICAL ASSESSMENT; Other: Questionnaires; Other: Thoracic-abdomino-pelvic scan or MRI
- Surveillance outside the trial (No Intervention)

INTERVENTIONS:
Drug: "FOLFIRI" cures — (Irinotecan 180 mg/m2, leucovorine 400mg/m2, 5FU bolus 400 mg/m2, 5FU continuous infusion 2400 mg/m2) every 14 days for 6 months or until disease progression on imaging
  Arms: Chemotherapy by FOLFIRI
Drug: Trifluridine cures — Trifluridine tipiracil 35 mg/m2 bid during 5 days/w on week 1 and 2 every 4 weeks, for 6 months or until disease progression on imaging
  Arms: Chemotherapy by Trifluridine tipiracil
Biological: BIOLOGICAL ASSESSMENT — blood sample ACE markers
  Arms: Chemotherapy by FOLFIRI; Chemotherapy by Trifluridine tipiracil; Surveillance inside the trial/control arm
Other: Questionnaires — Quality of life questionnaires (QLQ-C30 ; EQ-5D-5L ; GPAQ)
  Arms: Chemotherapy by FOLFIRI; Chemotherapy by Trifluridine tipiracil; Surveillance inside the trial/control arm
Other: Thoracic-abdomino-pelvic scan or MRI — Thoracic-abdomino-pelvic scan or MRI
  Arms: Chemotherapy by FOLFIRI; Chemotherapy by Trifluridine tipiracil; Surveillance inside the trial/control arm

SUMMARY:
Phase III multicentric, open-label, randomized study

The main objective is to assess the efficacy on time to disease recurrence (TTR) of treating minimal residual disease diagnosed by the presence of ctDNA after full treatment (surgery + chemotherapy) in stage III or high-risk stage II colon or upper rectum adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Fully resected stage III or high-risk stage II colon or upper rectum adenocarcinoma previously treated by standard adjuvant chemotherapy or peri-operative chemotherapy (FOLFOX or CAPOX) for either 3 or 6 months based on local multidisciplinary meeting, and on TNCD recommendations
* Positive ctDNA screening (methylation) and confirmation (NGS) on samples collected at the 3- or 6 months follow-up visit post-adjuvant chemotherapy
* Patients ≥ 18 years and ≤ 80 years (provided the score of the G8 geriatric questionnaire is >14 for patients 70 years or older)
* Subjects with WHO performance status < 2
* No documented disease using TAP CT-scanner and liver MRI in the case of contra-indication to dye contrast (or TEP-scanner may be also used in addition depending on physicians' choice and local availabilities).
* Adequate haematological function: with neutrophils ≥ 1,500 /mm3, platelet count ≥ 100,000/mm3, hemoglobin ≥ 9 g/dL (5,6 mmol/l)

Total bilirubin ≤ 1.5 x ULN (upper limit of normal) ASAT and ALAT ≤ 2.5 x ULN Alkaline phosphatase ≤ 2.5 x ULN Creatinine clearance ≥50 ml/min according MDRD (Modification of Diet in Renal Disease)

* Available tumor sample for NGS analysis
* Signed written informed consent obtained prior to any study specific procedures
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patients already treated with trifluridine tipiracil or irinotecan in the past 5 years
* Uncontrolled intercurrent illness
* Previous malignancies other than adequately treated in situ carcinoma of the uterine cervix or basal or squamous cell carcinoma of the skin, unless there has been a disease-free interval of at least 3 years
* Pregnant or breastfeeding women, women of childbearing age not having had a negative pregnancy test
* Any known specific contraindication or allergy to the treatments used in the study†
* Total or partial dihydropyrimidine dehydrogenase (DPD) deficiency (uracilemia > 16ng/ml)
* Known Gilbert's disease (UGT1A1*28 genotype)
* In case of concomitant use with St John's Wort related to irinotecan
* In case of bowel obstruction according related to irinotecan
* In case of recent concomitant treatment with brivudine, related to fluorouracil.
* Participation to another interventional study for postoperative therapy
* Persons deprived of liberty or under guardianship or incapable of giving consent
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1660 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The time to recurrence (TTR) | From date of randomization until the date of first documented progression or date of death from colorectal cancer
  The time to recurrence (TTR), in patients treated by FOLFIRI vs surveillance inside the study and in patients treated by Trifluridine Tipiracil vs surveillance inside the study. This TTR is defined as time from randomization to disease recurrence including locoregional or metastatic relapse, death with evidence of recurrence and death from CRC cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France